CLINICAL TRIAL: NCT06379360
Title: Maintenance Therapy of Hypomethylating Agent (HMA) in Favorable Risk Acute Myeloid Leukemia (AML) Patients: A Single Arm, Multi Center Clinical Trial
Brief Title: Maintenance Therapy of Hypomethylating Agent (HMA) in Favorable Risk Acute Myeloid Leukemia (AML) Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZAMLLRM01
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; favorable risk; azacitidine; decitabine; maintenance therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Decitabine

STUDY DESIGN:
Intervention Model Description: Apply hypomethylating agent, azacitidine or decitabine as maintenance therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMA maintenance therapy (Experimental): All enrolled patients received maintenance therapy consisting of azacitidine or decitabine.
  Interventions: Drug: Hypomethylating agent, Azacitidine or Decitabine

INTERVENTIONS:
Drug: Hypomethylating agent, Azacitidine or Decitabine — All enrolled patients received maintenance therapy consisting of Azacitidine (75mg/m2, subcutaneous injection, days 1-7) or Decitabine (20mg/m2, intravenous infusion, days 1-5), every three months as a cycle, for a maintenance therapy of 4-8 cycles.
  Other Names: Hypomethylating agent (HMA)

SUMMARY:
HMA maintenance therapy is expected to benefit overall survival (OS) and relapse free survival (RFS) in AML patients with favorable risk.

DETAILED DESCRIPTION:
Applying hypomethylating agents, azacitidine or decitabine as maintenance therapy in favorable-risk AML may prolong the remission duration and further improve their long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥16 years;
2. Patients diagnosed with AML and categorized into favorable-risk group according to European LeukemiaNet (ELN) 2022;
3. Patients achieved remission after induction therapy and finished at least 3 cycles of high-dose Aar-C based consolidation therapy, remaining in minimal residual disease (MRD) negative remission status (For NPM1-mutated and core binding factor acute myeloid leukemia (CBF-AML), MRD negative is defined as <2%, CEBPA-mutated AML, MRD negative is defined as <0.1%).
4. Patients not receiving hematopoietic stem cell transplantation prior to enrollment;
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
6. Expected survival time ≥ 3 months;
7. No serious heart, lung, liver or kidney disease;
8. Have the ability to understand and be willing to sign the informed consent form for this trial.

Exclusion Criteria:

1. Patients experienced hematologic relapse before recruitment.
2. Patients who are allergic to the study drug or drugs with similar chemical structures.
3. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception.
4. Active infection.
5. Active bleeding.
6. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment.
7. Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met.
8. Liver function abnormalities (total bilirubin > 1.5 times the upper limit of the normal range, Alanine Aminotransferase (ALT) / Aspartate Aminotransferase (AST) > 2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine > 1.5 times the upper limit of the normal value).
9. Patients with a history of clinically significant Corrected QT Interval (QTc) prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment.
10. Surgery on the main organs within the past six weeks.
11. Drug abuse or long-term alcohol abuse that would affect the evaluation results. Patients who have received organ transplants (excepting bone marrow transplantation).
12. Patients not suitable for the study according to the investigator's assessment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival (RFS) | 5 year
  It is measured from the date of entry into this trial to the date of hematologic relapse or death from any cause; subjects not known to have any of these events are censored on the date they were last examined.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 year
  It is measured from the date of entry into this trial to the date of death from any cause; subjects not known to have died at last follow-up are censored on the date they were last known to be alive.
Cumulative incidence of relapse (CIR) | 5 year
  CIR defined as from the time of recruitment to the study until the date of hematologic relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Li Xue, M.D., Principal Investigator — The First Affliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China